CLINICAL TRIAL: NCT02638896
Title: Efficacy and Safety of Etanercept Dose Reduction in Patients With Ankylosing Spondylitis
Brief Title: Dose Reduction of Etanercept in Patients With Ankylosing Spondylitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhixiang Huang (Other Government)
Responsible Party: Sponsor-Investigator, Zhixiang Huang, MD, Health and Family Planning Commission of Guangdong
Organization: Health and Family Planning Commission of Guangdong (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015117183344589
Record Dates: First submitted 2015-12-20; First posted 2015-12-23 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Etanercept; Sulfasalazine; Efficacy; Safety; dose; reduction
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept; Sulfasalazine; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose reduction arm (Experimental): AS patients who achieved remission will receive etanercept 50 mg subcutaneous injections every other weeks plus sulfasalazine (2g/d) oral administration till week24. Celecoxib will be the background therapy.
  Interventions: Drug: etanercept (Half-Dose); Drug: Sulfasalazine; Drug: Celecoxib
- Dose maintenance arm (Active Comparator): AS patients who achieved remission will receive etanercept 50 mg subcutaneous injections every weeks plus sulfasalazine (2g/d) oral administration till week24. Celecoxib will be the background therapy.
  Interventions: Drug: etanercept (Full-Dose); Drug: Sulfasalazine; Drug: Celecoxib
- Etanercept discontinuation arm (Other): AS patients who achieved remission will take sulfasalazine (2g/d) till week24. Celecoxib will be the background therapy.
  Interventions: Drug: Sulfasalazine; Drug: Celecoxib

INTERVENTIONS:
Drug: etanercept (Half-Dose) — AS patients who satisfied the criteria for disease remission (ASDAS<1.3) will be randomized to one of the three treatment arms. In the dose reduction arm, patients will receive etanercept 50 mg subcutaneous injections every other weeks .
  Other Names: Enbrel
  Arms: Dose reduction arm
Drug: etanercept (Full-Dose) — AS patients who satisfied the criteria for disease remission (ASDAS<1.3) will be randomized to one of the three treatment arms. In the dose maintenance arm, patients will receive etanercept 50 mg subcutaneous injections every weeks.
  Other Names: Enbrel
  Arms: Dose maintenance arm
Drug: Sulfasalazine — AS patients who satisfied the criteria for disease remission (ASDAS<1.3) will take sulfasalazine (2g/d) from week12 to week48.
  Other Names: Sulazine
Drug: Celecoxib — Celecoxib (0.4g/d) will be the background therapy.
  Other Names: Celebrex

SUMMARY:
The primary objective of this study is to evaluate the efficacy of safety of etanercept dose reduction combined with sulfasalazine in ankylosing spondylitis (AS) patients who have achieved a significant clinical response.

DETAILED DESCRIPTION:
This single-centre, open-labeled randomized study will evaluate the efficacy of safety of etanercept dose reduction combined with sulfasalazine in patients who achieved a significant clinical response. AS patients who meet the inclusion criteria will take celecoxib (0.4g/d) during the whole period of study. In the first period, all patients will be given etanercept 50 mg subcutaneous injections weekly from baseline to week12. In the second period, patients who satisfied the criteria for disease remission will be randomized to one of the following three treatment arms: (1) Dose reduction arm: Patients will receive etanercept 50 mg subcutaneous injections every other weeks plus sulfasalazine (2g/d) oral administration till week24. (2) Dose maintenance arm: Etanercept remains unchange from week12 to week24. (3) Etanercept discontinuation arm: Patients will be treated with sulfasalazine (2g/d) oral administration till week24. In the third period, all patients will take sulfasalazine (2g/d) till week 48. Ankylosing spondylitis disease activity score (ASDAS), erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), Bath ankylosing spondylitis functional index (BASFI), Bath ankylosing spondylitis metrology index (BASMI),Spondyloarthritis research consortium of Canada(SPARCC) score for the sacroiliac joint and adverse effect will be assessed in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 to 45 years of age.
2. Proven AS according to the modified New York criteria
3. Negative result of a pregnancy test in serum in screening visit and in urine in baseline visit, done in all women, except those surgically sterilized and those who have at least one year of menopause.
4. Sexually active women of childbearing potential must agree and commit to use a medically accepted form of contraception.
5. ASDAS score ≥2.1
6. Ability to reconstitute the drug and self-inject it or have a person who can do so.
7. Capability to understand and voluntarily give written informed consent that is signed and dated, before any specific procedure of the protocol is performed.
8. Ability to store injectable test article at 2º to 8º C.

Exclusion Criteria:

1. Pregnancy/lactation.
2. Previously exposure to murine or chimeric monoclonal antibodies.
3. Receipt of any live (attenuated) vaccines within 4 weeks before screening visit.
4. History of chronic or a recent serious infection.
5. History of tuberculosis within the last 3 years.
6. History of malignancy.
7. Significant concurrent medical diseases including uncompensated congestive heart failure, myocardial infarction within 12 months, stable or unstable angina pectoris, uncontrolled hypertension, severe pulmonary disease, history of human immunodeficiency virus (HIV) infection, central nervous system demyelinating events suggestive of multiple sclerosis.
8. Presence or history of confirmed blood dyscrasias.
9. History of any viral hepatitis within 1 year prior screening or history of any drug-induced liver injury at any time prior to screening.
10. Laboratory exclusions are: hemoglobin level < 8.5 mg/dl white blood cell count < 3.5×10e9/l, platelet count < 125 ×10e9/l, creatinine level > 175 mcmol/l, liver enzymes > 1.5 times the upper limit of normal or alkaline phosphatase > 2 times the upper limit of normal.
11. Participation in trials of other investigational medications within 30 days of entering the study.
12. Clinical examination showing significant abnormalities of clinical relevance.
13. Concomitant medication with disease-modifying anti-rheumatic drugs (DMARDs) or corticosteroids.
14. Hypersensitivity to any regent of study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change in ASDAS from baseline to week48. | Baseline, Week12, Week24, Week48
  ASDAS includes CRP (mg/L); Apart from the value of CRP, the four additional self-reported items (rated on 0-10 numerical rating scale [NRS]) included in this index are back pain, duration of morning stiffness, peripheral pain/swelling and patient global assessment of disease activity. The ASDAS scores are calculated as follows: ASDAS= (0.121×total back pain) + (0.110×subject global) + (0.073×peripheral pain/swelling) + (0.058×duration of morning stiffness) + (0.579×Ln(CRP+1)).

SECONDARY OUTCOMES:
Change in ESR from baseline to week48. | Baseline, Week12, Week24, Week48
  ESR is a laboratory test that provides a non-specific measure of inflammation. This test assesses the rate at which red blood cells fall in a test tube and is measured in mm/h. Normal range is 0 to 30 mm/h. A higher rate is consistent with inflammation.
Change in CRP from baseline to week48. | Baseline, Week12, Week24, Week48
  CRP is a marker of inflammation and measured in mg/L. A higher level is consistent with inflammation.
Change in BASFI from baseline to Week48. | Baseline, Week12, Week24, Week48
  BASFI is a validated self assessment tool that determines the degree of functional limitation in AS patients. Participants answered 10 questions, consisting of 8 specific questions regarding function in AS patients and 2 questions reflecting the participant's ability to cope with everyday life. Each question was answered on a 0-10 scale (0 being no problem and 10 being the worst problem), the sum of which (divided by 10) resulted in the BASFI score (0-10).
Change in BASMI from baseline to Week48. | Baseline, Week12, Week24, Week48
  BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10.
Change in SPARCC score for the sacroiliac joint from baseline to Week48. | Baseline, Week12, Week24, Week48
  SPARCC score for the sacroiliac joint was based on 6 consecutive coronal slices from posterior to anterior. Each joint was divided into 4 quadrants. Each quadrant was assigned a score of 0 = no lesion/1 = increased signal. For each slice, the score is increased by 1 for each joint that exhibits an intense signal in any quadrant. Also, for each slice, an additional score of 1 will be given for each joint that includes a lesion demonstrating continuous increased signal of a depth ≥1 cm from the articular surface. The maximum possible score is 72.
Percentage of participants with serious adverse events (SAEs) or adverse events (AEs) by co-morbidity from baseline to Week48. | Baseline, Week12, Week24, Week48
  Any untoward medical occurrence in a participant who received study regents was considered an AE, without regard to possibility of relationship. An AE resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a SAE: death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Tianwang Li, MD, Principal Investigator — Guangdong No.2 Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No